CLINICAL TRIAL: NCT01624103
Title: Influence of Anesthetic Volume on Comfort Score During US-SCB Placement in Elderly Patients
Brief Title: Comfort Score During Ultrasound Guided Supraclavicular Brachial Plexus Block Placement in Elderly Patients
Acronym: US-SCB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Šarić, Jadranka Pavičić, M.D. (Individual)
Responsible Party: Principal Investigator, Jadranka Pavičić Šarić, Principal Investigator, Clinical Hospital Merkur
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-000261-21
Record Dates: First submitted 2012-06-16; First posted 2012-06-20 (Estimated); Last update posted 2015-03-03 (Estimated); Status verified 2015-03

CONDITIONS: Arm Injuries; Wounds and Injuries
Keywords: Arm Injuries; Wounds and Injuries; Lidocaine; Levobupivacaine; Bupivacaine; Anesthetics; Central Nervous System Depressants; Physiological Effects of Drugs
MeSH Terms: conditions — Arm Injuries; Wounds and Injuries | interventions — Levobupivacaine; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Elderly (32 mL LA volume) (Experimental): Population over age of 65 undergoing upper limb surgery using US-SCB receiving 32 ml of LA (50:50 mixture of 0.5% levobupivacaine and 2% lidocaine).
  Interventions: Procedure: Upper limb surgery
- Elderly (20 ml LA volume) (Experimental): Population over age of 65 undergoing upper limb surgery using US-SCB receiving 20 ml of LA (50:50 mixture of 0.5% levobupivacaine and 2% lidocaine).
  Interventions: Procedure: Upper limb surgery

INTERVENTIONS:
Procedure: Upper limb surgery — Elderly patients undergoing upper limb surgery received 20 ml of LA volume (50:50 mixture of levobupivacaine 0.5% and lidocaine 2%) for US-SCB. An independent observer unaware of the LA volume recorded maximal pain intensity resulting from block placements, questioned the patients about possible unpleasant events linked to the performance of US-SCB and assessed patient's satisfaction.
  Other Names: Levobupivacaine; Lidocaine; Chirocaine; Xilocaine
  Arms: Elderly (20 ml LA volume)
Procedure: Upper limb surgery — Elderly patients undergoing upper limb surgery received 32 ml of LA volume (50:50 mixture of levobupivacaine 0.5% and lidocaine 2%) for US-SCB. An independent observer unaware of the LA volume recorded maximal pain intensity resulting from block placements, questioned the patients about possible unpleasant events linked to the performance of US-SCB and assessed patient's satisfaction.
  Other Names: Levobupivacaine; Lidocaine; Chirocaine; Xilocaine
  Arms: Elderly (32 mL LA volume)

SUMMARY:
Results from our preliminary study accepted as e-poster presentation on ESRA (Bordeaux, September 2012.) showed significant difference in Comfort Score during Ultrasound Guided Supraclavicular Brachial Plexus block (US-SCB) between young and elderly population. However, it is unknown whether the difference in Comfort score (1) was associated with reduction of local anesthetic (LA) volume in elderly or it is attributed to elderly population by itself. The aim of the study is to compare the Comfort score during US-SCB placement in elderly patients undergoing upper limb surgery performed with two different volumes of local anesthetics (20 ml vs 32 ml).

DETAILED DESCRIPTION:
Involutional changes of brachial plexus in elderly, assessed by measuring the cross-sectional area (CSA) of brachial plexus at the first rib, allowed a 35% reduction of LA volume for an effective US-SCB in comparison with the younger patients (2). Ultrasound-guided regional anesthesia becomes an increasingly popular technique and its performance must be as comfortable as possible. Therefore, Comfort score during block placement is extremely important. Comfort Score is consisted of maximum pain intensity (VAS), the satisfaction of the patient and the number of unpleasant events declared by the patients. It is calculated as the sum of each criterion, which was attributed a value of 0 or 1: VAS(<or=30/100, 1; >30/100, 0), number of unpleasant events (0, 1; >or=1, 0) and satisfaction (satisfied or very satisfied, 1; acceptable or unsatisfied, 0). Comfort score of 3 or 2 is considered as comfortable while score 1 or 0 as uncomfortable block placement.

ELIGIBILITY:
Inclusion Criteria:

* age over 65 years (Elderly group)
* upper limb surgery

Exclusion Criteria:

* refusal of regional anesthesia
* any neurologic or neuromuscular disease
* clinical signs of cutaneous infection at the site of needle insertion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Comfort Score | Up to average 20 min
  An independent observer unaware of the administered LA volume assessed Comfort score by evaluating maximal pain intensity resulting from block placement using a 100-mm visual analogue scale (VAS: 0, no pain-100, maximum or worst imaginable) as well as by recording any unpleasant event during block placement and by recording patient satisfaction using a four-point scale (unsatisfied, acceptable, satisfied and very satisfied).

SECONDARY OUTCOMES:
Block Placement Time | Up to average 20 minutes
  Block placement time was measured as the time elapsing between needle insertion and to last removal of the needle from the patient's neck.

CONTACTS AND LOCATIONS:
Overall Officials: Matea Bogdanović Dvorščak, MD, Study Chair — Clinical Hospital Merkur, Department of Anesthesiology and Intensive Care
Locations (1):
- Clinical Hospital Merkur, Zagreb, City of Zagreb, Croatia

REFERENCES:
- [Background] Bloc S, Mercadal L, Garnier T, Komly B, Leclerc P, Morel B, Ecoffey C, Dhonneur G. Comfort of the patient during axillary blocks placement: a randomized comparison of the neurostimulation and the ultrasound guidance techniques. Eur J Anaesthesiol. 2010 Jul;27(7):628-33. doi: 10.1097/EJA.0b013e328333fc0a. PMID 20299995
- [Background] Tomulic K, Pavicic Saric J, Acan I.Effect of age on anaesthetic volume for ultrasound guided supraclavicular brachial plexus block: 8AP2-8 European Journal of Anaesthesiology 28:113,2011